CLINICAL TRIAL: NCT03464500
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy of AMAZ-02 on Muscle Function in Otherwise Healthy Middle-aged, Overweight and Inactive Individuals
Brief Title: AMAZ-02 Effect on Exercise ToLerance in Healthy, Overweight Middle Aged Subjects (ATLAS Trial)
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18AMHA / 17.02.AMZ
Record Dates: First submitted 2018-02-05; First posted 2018-03-14 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2019-10

CONDITIONS: Muscle Function, Mitochondrial Function; Overweight; Healthy Aging
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mitopure 500mg (Active Comparator)
  Interventions: Dietary Supplement: Mitopure 500mg
- Mitopure 1000mg (Active Comparator)
  Interventions: Dietary Supplement: Mitopure 1000mg
- Placebo (Active Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mitopure 500mg — Mitopure containing softgels
  Arms: Mitopure 500mg
Dietary Supplement: Mitopure 1000mg — Mitopure containing softgels
  Arms: Mitopure 1000mg
Dietary Supplement: Placebo — Placebo containing softgels
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled study enrolling 90 healthy, overweight, middle aged subjects (30 placebo, 30 low dose and 30 high dose AMAZ-02 intervention), 40-65 years of age, who are otherwise healthy. AMAZ-02, a food derived ingredient, will be given as a daily oral dose for 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females 40 to 65 years of age, inclusive
2. Subjects who have not participated within the last 1 year in clinical trials focused on improving muscle function and physical performance
3. Female participant is not of child bearing potential, defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) or,

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner (shown successful as per appropriate follow-up)
4. Body mass index (BMI) between 25.0 and 34.9 kg/m2, inclusive
5. Agree to avoid exercising 24 hours prior to study visits and maintain low physical activity status for the duration of the trial
6. Agree to refrain from consumption of pomegranate juice and walnuts from 2 weeks prior to baseline and through the study period
7. Agree to limit consumption of raspberries, strawberries and cloudberries from 2 weeks prior to baseline and through the study period
8. Agree to refrain from using NSAIDs for 7-days prior to and following muscle sample collection
9. Good general health to perform exercise testing safely, as determined by the Qualified Investigator based on medical history, physical examination, ECG and laboratory results
10. Low VO2max defined as <35 ml/kg/min for males and <31 ml/kg/min for females as assessed by a submaximal cycle ergometer test
11. Comprehension of the nature and purpose of the study including possible risks and side effects, and ability to communicate in person and by telephone in a manner that allows all protocol procedures to be carried out safely and reliably in the opinion of the investigative site staff
12. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Smokers or ex-smokers within the past 1 year from screening, including use of vaporizers or e-cigarettes
3. Participation in another clinical study or receipt of an investigational drug within 60 days of the screening visit
4. Blood donation within 1 month of baseline, as well as planned donation 1 month after end of study.
5. Recent history (within the last 2 years) of alcohol or other substance abuse
6. Use of medicinal marijuana.
7. Unable to swallow capsules
8. Regular participation in a structured exercise program with physical activity levels in Category 2 or higher defined as 20 min vigorous activity 3-times per week, moderate activity for 30 min 5 days per week or more
9. Inability to abstain from intensive muscular effort
10. Individuals who have engaged in 1 hour or more per week of resistance training in the past 3 months.
11. Currently experiencing any medical condition that interferes with the ability to undergo physical strength testing during the study
12. Recent participation in a weight loss diet, or loss >5% of total body weight within 3 months of randomization
13. Clinically significant abnormal laboratory results at screening
14. Allergy or sensitivity to test product ingredients (or closely related compounds)
15. Allergy to anesthetic (Xylocaine, lidocaine)
16. Soy allergy
17. Inability to abstain from the consumption of pomegranate juice or walnuts
18. Inability to abstain from frequent consumption of raspberries, strawberries or cloudberries
19. Excessive consumption of beverages containing xanthine bases (>4 cups per day) such as coffee, tea, and cola
20. Use of NHPs for the purposes of muscle building or function. Use of other NHPs must have been on a stable dosing regimen for at least a month prior to baseline and must maintain their current dosing regimen throughout the trial and must not begin taking any new NHPs throughout the trial; if the subject wishes to stop taking the NHP prior to beginning the trial they must do so at least 2 weeks prior to randomization.
21. History of or current diagnosis of bleeding/blood disorder
22. Use of oral anticoagulants (blood thinners), New Oral Anticoagulants (NOAC) or antiplatelet agents.
23. Use of NSAID medications within one week before or after the needle muscle biopsy procedures.
24. Use of steroid medications, current/recent (3 months) history of anabolic steroid, corticosteroid or estrogen use.
25. Use of statins
26. Use of thyroid medications.
27. Asthma that has not been controlled with a stable regimen for a minimum of a year, or Asthma requiring the use of certain medications.
28. Diagnosis of COPD
29. Chronic myalgia, fibromyalgia or conditions characterized by regular muscle pain
30. Metal fixation plates or screws from a previous surgery
31. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may confound the study outcomes (i.e. terminal illnesses)
32. Diagnosis of active cardiac or peripheral vascular disease
33. SBP/DBP ≥150/95 mmHg without the use of hypertension medications, or SBP/DBP >140/90 mmHg with the use of hypertension medications.
34. Diagnosed hyperlipidemia
35. Renal or hepatic impairment or disease
36. Any major diseases of the gastrointestinal, pulmonary or endocrine systems
37. Type I and Type II diabetes
38. Autoimmune disease or immuno-compromised (i.e. HIV positive, use of anti-rejection medication, rheumatoid arthritis, Hepatitis B/C positive)
39. Diagnosis of chronic infectious disease
40. Diagnosis of phenylketonuria
41. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Participants with cancer in full remission for more than five years after diagnosis are acceptable if approved by QI.
42. Significant neurological or psychiatric illness, including, but not limited to, Parkinson's disease and bipolar disorder as assessed by QI.
43. History of seizures
44. Individuals who are cognitively impaired and/or who are unable to give informed consent
45. Any other condition which in the qualified investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in exercise tolerance as assessed by power output on the cycle ergometer from baseline to day 120 between AMAZ-02 groups and placebo | 4 months

SECONDARY OUTCOMES:
Change in exercise tolerance as assessed by power output on the cycle ergometer from baseline to day 60 between AMAZ-02 groups and placebo | 2 months
Change in exercise tolerance as assessed by time to fatigue on the cycle ergometer from baseline to day 60 and from baseline to day 120 between AMAZ-02 groups and placebo | 2, 4 months
Change in handgrip strength of the non-dominant hand as assessed by Jamar dynamometry from baseline to day 120 between AMAZ-02 groups and placebo | 4 months
Change in isokinetic lower body muscle strength as assessed by the Biodex isokinetic dynamometer from baseline to day 120 between AMAZ-02 groups and placebo | 4 months
Change in physical performance on the cycle ergometry defined as the time to reach 85% of maximum heart rate from baseline to days 60 and from baseline to day 120 between AMAZ-02 groups and placebo | 2, 4 months
Change in distance walked in the 6-minute walk test as a measure of aerobic endurance from baseline to day 120 between AMAZ-02 groups and placebo | 4 months
Change in gait speed from baseline to day 120 between AMAZ-02 groups and placebo as derived from the 6-minute walk test | 4 months
Change in the 30-second chair stand test from baseline to day 120 between AMAZ-02 groups and placebo | 4 months
Change from baseline to days 60 and from baseline to day 120 between AMAZ-02 groups and placebo in participant's quality of life as assessed by the 36-item short form (SF-36) questionnaire | 4 months
Change from baseline to days 60 and from baseline to day 120 between AMAZ-02 groups and placebo in participant's perceived exertion during exercise testing as assessed by the Borg Rating of Perceived Exertion Scale (Scale from 6-20) | 2, 4 months
Change from baseline to days 60 and 120 between AMAZ-02 groups and placebo in participant' resting energy expenditure in Kcal/ day via the Cardiocoach CO2 system | 2, 4 months
Change in 3-day food records reviewed at baseline and days 60 and 120 | 2, 4 months
Change from baseline to day 60 and from baseline to day 120 in serum lipid profile, insulin, and HbA1C between AMAZ-02 groups and placebo | 2, 4 months
Change in lean body mass as assessed by dual X-ray absorptiometry (DXA) from baseline to day 120 between AMAZ-02 groups and placebo | 4 months
Change in acylcarnitine profile in plasma via Metabolomics assessments from baseline to day 60, and from baseline to day 120 between AMAZ-02 groups and placebo | 2, 4 months
Change in plasma muscle function biomarkers (myostatin, follistatin, inflammatory cytokines and mitokines) from baseline to day 60 and from baseline to day 120 between AMAZ-02 groups and placebo | 2, 4 months
Change in in vivo mitochondrial gene expression from baseline to day 120 between AMAZ-02 groups and placebo as assessed via microarray performed on muscle biopsy | 4 months
Change in the gut microbial diversity at baseline and at day 120 between AMAZ-02 groups and placebo assessed via 16s RNA sequencing performed on fecal samples | 4 months
The change in the international physical activity questionnaire score (IPAQ) from baseline to day 120 between AMAZ-02 500mg/d and 1000mg/d and placebo. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mal Evans, PhD, Study Director — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada

REFERENCES:
- [Background] Singh A, D'Amico D, Andreux PA, Fouassier AM, Blanco-Bose W, Evans M, Aebischer P, Auwerx J, Rinsch C. Urolithin A improves muscle strength, exercise performance, and biomarkers of mitochondrial health in a randomized trial in middle-aged adults. Cell Rep Med. 2022 May 17;3(5):100633. doi: 10.1016/j.xcrm.2022.100633. PMID 35584623
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35584623/